CLINICAL TRIAL: NCT04448899
Title: Effects of Ivabradine on Neopterin and NT-Pro BNP in Patients With Congestive Heart Failure
Brief Title: Ivabradine in Patients With Congestive Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Principal Investigator, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ivabradine in CHF
Record Dates: First submitted 2020-06-24; First posted 2020-06-26 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivabradine (Active Comparator): Patients administered Ivabradine 5 mg twice daily and doses (2.5, 5, 7.5 mg) were to be adjusted upwards or downwards at every visit according to HR at rest and tolerability.
  Patients were followed up after 1 week of initiation of ivabradine therapy then monthly till the end of the study.
  Interventions: Drug: Ivabradine Oral Tablet
- Control (Placebo Comparator): Patients administered a placebo twice daily. Patients were followed up after 1 week of initiation of the study then monthly till the end of the study.
  Interventions: Drug: Blacebo plus standard treatment

INTERVENTIONS:
Drug: Ivabradine Oral Tablet — Ivabradine 5 mg twice daily and doses (2.5, 5, 7.5 mg) were to be adjusted upwards or downwards at every visit according to HR at rest and tolerability plus their standard treatment.
  Other Names: Procoralan 5 mg film-coated tablets
  Arms: Ivabradine
Drug: Blacebo plus standard treatment — Blacebo plus standard treatment
  Arms: Control

SUMMARY:
The aim of this study is to assess the efficacy of Ivabradine therapy in patients with congestive heart failure using the cardiac biomarkers NT-Pro BNP and Neopterin.

DETAILED DESCRIPTION:
* Approval will be obtained from Research Ethics Committee of Faculty of Pharmacy, Damanhour University
* All participants have agreed to take part in this clinical study and provide informed consent
* A 3 months, prospective interventional study.
* Sixty ambulatory, clinically stable symptomatic patients with systolic chronic HF (≥ 4 weeks), on optimized standard medical therapy were consecutively included and randomly allocated to the ivabradine group (n=30) and non-ivabradine group (n=30).
* The baseline evaluation comprised physical examination, NYHA class, 12-lead electrocardi¬ography (ECG), Echocardiography, blood sampling for laboratory measurements, including NT-Pro BNP and Neopterin.
* Patients in the Ivabradine group were administered Ivabradine 5 mg twice daily and doses (2.5, 5, 7.5 mg) were to be adjusted upwards or downwards at every visit according to HR at rest and tolerability.
* Patients were followed up after 1 week of initiation of ivabradine therapy then monthly till the end of the study.
* Peripheral venous blood samples were drawn between 8 and 9 am after a 30-min rest in the supine position. Serum samples were frozen at -80°C until assay.
* Levels of NT-Pro BNP and Neopterin were detected using ELISA kits as prescribed by manufacturer.
* Statistical tests appropriate to the study will be conducted to evaluate significance of results
* Results, conclusion, discussion and recommendations will be given

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic HF, on optimized medical therapy according to European Society of Cardiol¬ogy guidelines, with LV ejection fraction (LVEF) < 35% according to the Simpson method, New York Heart Association (NYHA) class II-III, and sinus rhythm and resting HR > 70/min were eligible for inclusion in the study.

Exclusion Criteria:

* acute decompen¬sation (acute coronary syndromes and acute HF);
* hemodynamically significant valve disease;
* cer¬ebrovascular events during the previous 6 months;
* dysfunctional prosthetic heart valve;
* obstructive or non-obstructive cardiomyopathy; uncorrected congenital heart disease; active myocarditis;
* a his¬tory of resuscitation from sudden death; an absence of stable sinus rhythm, severe arrhythmias; HR < 60 bpm; sick sinus syndrome; second-degree and third-degree atrioventricular block;
* severe obesity (body mass index > 36 kg/m²);
* established or sus¬pected pulmonary diseases (vital capacity < 80% or forced expiratory volume in 1 s < 80% of age spe¬cific and sex-specific reference values);
* hemoglobin ≤ 11 g/dL;
* treatment with non-dihydropyridine calcium-channel blockers, class I antiarrhythmic agents, strong inhibitors of cytochrome P450-3A4, or QT interval-prolonging medications;
* acute and chronic kidney failure;
* pregnancy; hypo- and hy¬perthyroidism or acute infections.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
NT-Pro BNP | three months
  Serum BNP (pg/ml)
Neopterin | three months
  Serum Neopterin (nmol/L)

SECONDARY OUTCOMES:
Heart Rate | Three Months
  Heart Rate (Beat/Minute)

CONTACTS AND LOCATIONS:
Overall Officials: Rehab Werida, Lecturer, Study Director — Damanhour University, Faculty of Pharmacy; Jayda M Dogheim, B. Pharm, Principal Investigator — Alexandria University
Locations (1):
- Tanta University Hospital, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Komajda M, Tavazzi L, Francq BG, Bohm M, Borer JS, Ford I, Swedberg K; SHIFT Investigators. Efficacy and safety of ivabradine in patients with chronic systolic heart failure and diabetes: an analysis from the SHIFT trial. Eur J Heart Fail. 2015 Dec;17(12):1294-301. doi: 10.1002/ejhf.347. Epub 2015 Sep 16. PMID 26377342
- [Result] Tavazzi L, Swedberg K, Komajda M, Bohm M, Borer JS, Lainscak M, Ford I; SHIFT Investigators. Efficacy and safety of ivabradine in chronic heart failure across the age spectrum: insights from the SHIFT study. Eur J Heart Fail. 2013 Nov;15(11):1296-303. doi: 10.1093/eurjhf/hft102. Epub 2013 Jun 26. PMID 23803951
- [Result] Sasaki T, Takeishi Y, Suzuki S, Niizeki T, Kitahara T, Katoh S, Ishino M, Shishido T, Watanabe T, Kubota I. High serum level of neopterin is a risk factor of patients with heart failure. Int J Cardiol. 2010 Nov 19;145(2):318. doi: 10.1016/j.ijcard.2009.11.042. Epub 2010 Jan 6. PMID 20051294
- [Result] Richards M, Troughton RW. NT-proBNP in heart failure: therapy decisions and monitoring. Eur J Heart Fail. 2004 Mar 15;6(3):351-4. doi: 10.1016/j.ejheart.2004.01.003. PMID 14987587